CLINICAL TRIAL: NCT00799656
Title: Efficacy and Safety of Oral Ataciguat (HMR1766) 200 mg Administered Once Daily for 28 Days on Pain Reduction in Patients With Neuropathic Pain. A Randomized, Double-blind, Placebo-controlled, Cross-over Study
Brief Title: Efficacy and Safety Study of Ataciguat Versus Placebo in Patients With Neuropathic Pain
Acronym: SERENEATI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: DFI10569; EudraCT 2008-001518-26
Record Dates: First submitted 2008-11-27; First posted 2008-12-01 (Estimated); Last update posted 2011-04-01 (Estimated); Status verified 2011-03

CONDITIONS: Pain
Keywords: Diabetic neuropathy; painful pain; postoperative
MeSH Terms: conditions — Pain; Diabetic Neuropathies | interventions — 5-chloro-2-(5-chlorothiophene-2-sulfonylamino)-N-(4-(morpholine-4-sulfonyl)phenyl)benzamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): First period: Ataciguat - Second period: Placebo
  Interventions: Drug: ataciguat (HMR1766); Drug: placebo
- 2 (Experimental): First period: Placebo - Second period: Ataciguat
  Interventions: Drug: ataciguat (HMR1766); Drug: placebo

INTERVENTIONS:
Drug: ataciguat (HMR1766) — oral administration 200mg once daily for 28 days
Drug: placebo — oral administration once daily for 28 days

SUMMARY:
The primary objective of this study is to assess the efficacy of ataciguat versus placebo in reducing pain intensity in patients with neuropathic pain.

The secondary objective is to assess the safety and tolerability of ataciguat versus placebo.

DETAILED DESCRIPTION:
This study consists of two consecutive 28 day treatment periods which are separated by a 2 week medication free period and a safety follow-up period of 2 weeks after the second treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic neuropathic pain due to diabetic polyneuropathy or a nerve lesion following surgery. The pain must be present for more than 3 months.

Exclusion Criteria:

* Presence or history of cancer within the past five years
* Patients with a history of HIV infection
* Patients with active hepatitis B or C
* Patients with any pain other than the neuropathic pain of greater or equal severity
* Patients with a diabetes mellitus for less than 6 months

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-11; Primary Completion 2009-06 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Change in average daily pain intensity | after 28-days treatment

SECONDARY OUTCOMES:
Responder rate | after 28-days treatment
Rescue medication intake | during 28-days treatment
Change in Neuropathic Pain Symptom Inventory (NPSI) | after 28-days treatment

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Goerg Kress, Professor, Principal Investigator — Medizinische Universität / AKH Wien - Währinger Gürtel 18-20 - A-1090 Wien
Locations (3):
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Bucharest, Romania